CLINICAL TRIAL: NCT06265519
Title: The Association of Urinary BDNF and NGF With Lower Urinary System Parameters in Patients With Bladder Outlet Obstruction Secondary to Benign Prostate Hyperplasia
Brief Title: Association of Urine BDNF and NGF With Lower Urinary System Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MAR.UAD.008
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia With Outflow Obstruction; Lower Urinary Tract Obstructive Syndrome

STUDY DESIGN:
Masking Description: 0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients before surgery (Active Comparator): Men between the ages of 50 and 80 diagnosed with BPH before surgery
  Interventions: Procedure: Holmium laser enucleation of the prostate
- Patients after surgery (Active Comparator): Men between the ages of 50 and 80 diagnosed with BPH after surgery
  Interventions: Procedure: Holmium laser enucleation of the prostate
- Healthy (No Intervention): Men between the ages of 50-80 years without lower urinary tract disease

INTERVENTIONS:
Procedure: Holmium laser enucleation of the prostate — Holmium laser enucleation of the prostate is a minimally invasive procedure that uses pulses of laser beam to remove tissue from the inside of the prostate, which surrounds the urethra (the tube leading from the bladder to the urinary opening) in patients with BPH
  Arms: Patients after surgery; Patients before surgery

SUMMARY:
Histologically, BPH is a benign proliferative process involving both epithelial and stromal elements and is characterised by progressive enlargement of the prostate. Symptom complex including increased frequency of urination, sudden feeling of urge to urinate, nocturia, difficulty in urinating, feeling of incomplete emptying of the bladder, decreased flow rate and intermittent urination are called lower urinary tract symptoms (LUTS). The most important cause of LUTS in men is BPH. Many structural and physiological changes occur in the lower urinary system with bladder outlet obstruction. Detrusor hypertrophy and bladder hyperactivity may occur due to bladder outlet obstruction. Although the density of afferent and efferent nerves in the bladder decreases after urethral obstruction, enlargement of their trunks indicates that changes occur in these nerves. In addition, changes also occur in the neural pathways of the central nervous system following lower urinary tract obstruction. Nerve growth factor (NGF) and brain derived neurotropin factor (BDNF) are trophic proteins that act as retrograde messengers between peripheral effector tissue and the nerves that innervate it. In peripheral tissues, the source of NGF and BDNF is presumed to be the target tissues innervated by nerves. Smooth muscle cells, fibroblasts, astrocytes and other cells synthesise NGF and BDNF in culture medium. Many potential stimuli that increase NGF in the lower urinary system have been identified. These are denervation, inflammation and mechanical tension. This information has led to the idea that autonomic innervation changes in the bladder may be related with changing NGF levels. Altered afferent and adrenergic innervation in the obstructed bladder increases the possibility that NGF plays an important role in this neural growth because this type of nerves are highly sensitive to this neurotrophin.

In this study, we investigated NGF ve BDNF levels in urine samples obtained before surgery (Transurethral Prostate Resection, Prostate Enucleation with Holmium Laser and Prostate Enucleation with Thulium Fibre Laser) and after removal of obstruction in patients with bladder outlet obstruction secondary to benign prostatic enlargement using ELISA method, We aimed to determine the role of NGF and BDNF in bladder outlet obstruction and bladder changes secondary to obstruction by comparing with control patients without obstruction.

DETAILED DESCRIPTION:
As the demographic structure of societies changes, benign prostatic hyperplasia (BPH) is one of the most important health problems for older men, especially in developed countries. Histologically, BPH is a benign proliferative process involving both epithelial and stromal elements and is characterised by progressive enlargement of the prostate. BPH is a lifelong chronic disease with an incidence of approximately 8% in men aged 31-40 years, which increases rapidly with age and reaches 90% in the 9th decade. Symptom complex including increased frequency of urination, sudden feeling of urge to urinate, nocturia, difficulty in urinating, feeling of incomplete emptying of the bladder, decreased flow rate and intermittent urination are called lower urinary tract symptoms (LUTS). The most important cause of LUTS in men is BPH. Many structural and physiological changes occur in the lower urinary system with bladder outlet obstruction. Detrusor hypertrophy and bladder hyperactivity may occur due to bladder outlet obstruction. Although the density of afferent and efferent nerves in the bladder decreases after urethral obstruction, enlargement of their trunks indicates that changes occur in these nerves.

In addition, changes also occur in the neural pathways of the central nervous system following lower urinary tract obstruction. Nerve growth factor (NGF) and brain derived neurotropin factor (BDNF) are trophic proteins that act as retrograde messengers between peripheral effector tissue and the nerves that innervate it. In peripheral tissues, the source of NGF and BDNF is presumed to be the target tissues innervated by nerves. Smooth muscle cells, fibroblasts, astrocytes and other cells synthesise NGF and BDNF in culture medium. NGF is required for survival, development and neurotransmitter synthesis regulation of dorsal root ganglion and sympathetic cells in embryonic and postnatal life . NGF receptor contains two subunits; the low affinity subunit is called p75 and the high affinity tyrosine kinase subunit is called tyrosine kinase A which is responsible for the growth and survival effects of NGF. Many potential stimuli that increase NGF in the lower urinary system have been identified. These are denervation, inflammation and mechanical tension. This information has led to the idea that autonomic innervation changes in the bladder may be related with changing NGF levels. Altered afferent and adrenergic innervation in the obstructed bladder increases the possibility that NGF plays an important role in this neural growth because this type of nerves are highly sensitive to this neurotrophin. Clinical and experimental data have shown a relationship between urinary NGF and overactive bladder. Overactive bladder (OAB) is a complex of uncomfortable symptoms accompanied by a feeling of urgency, frequent urination and nocturia, with or without urge incontinence. Overactive bladder is thought to occur as a result of an inflammatory process occurring in the bladder. The reason for this is shown as high levels of inflammation mediators in bladder biopsies and urine of OAB patients. NGF, which is one of the inflammation mediators, was found to be high in OAB patients in studies and it was observed that NGF level decreased after antimuscarinic treatment or botulinum neurotoxin injection.

In this study, we investigated NGF ve BDNF levels in urine samples obtained before surgery (Transurethral Prostate Resection, Prostate Enucleation with Holmium Laser and Prostate Enucleation with Thulium Fibre Laser) and after removal of obstruction in patients with bladder outlet obstruction secondary to benign prostatic enlargement using ELISA method, We aimed to determine the role of NGF and BDNF in bladder outlet obstruction and bladder changes secondary to obstruction by comparing with control patients without obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years Male
2. Patients with bladder outlet obstruction secondary to benign prostate hyperplasia

Exclusion Criteria:

1. Known neurological disease
2. Diabetes
3. Urinary tract infection
4. Previous prostate surgery
5. Spinal Cord Trauma

7-Bladder stone 8-Cerebrovascular disease 9-Chronic Renal Failure 10-Ureteral stenosis

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Uroflowmetry | 1 year
  Uroflowmetry is a test that measures the volume of urine released from the body, the speed with which it is released, and how long the release takes.

SECONDARY OUTCOMES:
International prostate symptom score | 1 year
  International prostate symptom score

OTHER OUTCOMES:
Urodynamic | Before surgery
  Urodynamic testing is any procedure that looks at how well parts of the lower urinary tract-the bladder, sphincters, and urethra-work to store and release urine.

CONTACTS AND LOCATIONS:
Overall Officials: Tufan Tarcan, Prof. Dr., Study Director — Marmara University; Çağrı Akın Şekerci, Assoc. Prof., Study Director — Marmara University; Banu İşbilen Başok, Prof. Dr., Study Director — Dr. Behçet Uz Children's Hospital; Kader Ada Doğan, MD, Study Director — Marmara University
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No